CLINICAL TRIAL: NCT00920686
Title: A Phase 2 Study of the Safety and Effectiveness of a Single Oral Dose of NXN 188 for the Treatment of Moderate to Severe Migraine Headache With Aura
Brief Title: Study of NXN 188 for the Treatment of Migraine With Aura
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeurAxon Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NXN-188-203
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-07

CONDITIONS: Migraine With Aura
Keywords: Migraine; aura
MeSH Terms: conditions — Migraine with Aura; Migraine Disorders; Epilepsy | interventions — Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NXN-188 (Experimental): NXN-188, 600 mg, PRN
  Interventions: Drug: NXN-188
- sumatriptan succinate 100 mg (Active Comparator): Sumatriptan, 100 mg, PRN
  Interventions: Drug: sumatriptan succinate
- placebo (Placebo Comparator): matching, PRN
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NXN-188 — NXN-188 hard gelatin capsules, 600 mg administered as three 200 mg capsules
  Other Names: NXN-188 dihydrochloride
  Arms: NXN-188
Drug: placebo — administered as 3 placebo hard gelatin capsules
  Other Names: placebo capsules
  Arms: placebo
Drug: sumatriptan succinate — administered in a hard gelatin capsule with 2 capsules of placebo
  Arms: sumatriptan succinate 100 mg

SUMMARY:
NXN-188 Dihydrochloride is being developed as an immediate release oral product for the treatment of acute migraine. This study is being conducted to evaluate NXN-188 in subjects with a migraine history of aura.

DETAILED DESCRIPTION:
This was a multicenter, double-blind, parallel group, active and placebo-controlled, three arm study of a single oral dose of NXN-188 for the treatment of acute migraine headache with aura.

After study eligibility was confirmed, subjects were randomized to NXN-188 600 mg, sumatriptan 100 mg, or placebo in a 1:1:1 ratio. Subjects left the clinic to self-administer the treatment at home at the onset of moderate to severe headache in a suitable dosing environment.

Treatment was not to exceed 42 days from Randomization. If the subject did not have a headache within 42 days of randomization (s)he did not take the study medication and returned it to the site. If the subject experienced a qualifying headache (s)he recorded the symptoms in a diary, dosed with the study drug, and called the IVRS to record assessments all adverse events and to report dosing. If the study drug provided insufficient relief 2 hours post dosing (s)he was permitted to use non-triptan rescue medication recommended by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female migraineurs between 18 and 65 years old.
2. Subjects must have a headache history of migraine with aura as defined by:

   * Aura consisting of at least one of the following, but no muscle weakness or paralysis:

     * Fully reversible visual symptoms
     * Fully reversible sensory symptoms
     * Fully reversible dysphasia
   * Aura has at least two of the following characteristics:

     * Visual symptoms affecting only one side of the field of vision and/or sensory symptoms affecting only one side of the body
     * At least one aura symptom that develops gradually over more than 5 minutes and/or different aura symptoms occur in succession over more than 5 minutes
     * Each symptom lasts from 5-60 minutes
   * Headache begins during the aura or follows aura within 60 minutes
   * Headache not attributable to another disorder
3. Migraine pain following aura in at least 75% of occurrences
4. Headache frequency of at least 1 migraine attack (with or without aura) per month for the past 3 months but not more than 8 migraines in any 30 day period. Subjects must have at least 1 migraine headache with aura per month

   • Each migraine attack should last at least 4 hours (without treatment) and not longer than 72 hours.
5. At the time of the study migraine, prior to dosing with study medication, the headache severity, as judged and documented by the subject, is either moderate or severe (on a 4-point categorical scale)
6. Body mass index (BMI) range of 18 to 35
7. The subject is in general good health.

   • ALT cannot be above 1.5x upper limit of normal; creatinine and urea must be within normal limits
8. Speak, read, and understand English, French, or Spanish sufficiently to understand the nature of the study, to provide written informed consent, and complete all study assessments
9. The subject is willing and able to comply with all testing requirements defined in the protocol
10. All females will avoid pregnancy at least 10 days before randomization, and up until 3 months after dosing.
11. All subjects/partners must use a double-barrier method of birth control during the study and for 3 months after dosing.

Exclusion Criteria:

1. A diagnosis of headaches that is not consistent with migraine with aura.
2. Presence of any risk factors that would preclude the use of triptans:
3. Known allergy or hypersensitivity to triptans or history of any serious side effect with a triptan which would preclude further dosing with a triptan
4. Presence of any clinically significant condition that would preclude study participation, as evaluated by the investigator
5. Pregnancy or lactation
6. History of significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, rheumatologic, autoimmune, or metabolic disease
7. Use of the following if taken for migraine prevention:

   * Cardiovascular drugs (acceptable if reason for use is for treatment of cardiovascular disease and the subject has been on a stable dose for 3 months)
   * Valproate, topiramate, cyproheptadine, montelukast, or botulinum toxin.
8. Use of monoamine oxidase inhibitors within 30 days of randomization
9. Initiation of therapy with SSRIs or SNRIs for depression or other approved indication within 90 days of randomization (subjects on stable dose for >3 months for treatment of depression or other approved indication may be included)
10. Are known to or suspected to be currently abusing alcohol or drugs, or have a history (within the past 12 months) of active alcohol or drug abuse
11. Participation in another drug or biologic study within 30 days of randomization into this study or during participation in this study
12. Subjects who are unable or unwilling, in the opinion of the Investigator, to comply with all study procedures and cooperate fully with study center staff

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Boudreau, MD, Principal Investigator — Hopital Notre-Dame Du Chum, Montreal
Locations (16):
- United States (16):
  - C. Philip O'Carrroll, MD, Inc., Newport Beach, California
  - The Research Center of Southern California, LLC, Oceanside, California
  - San Francisco Headache Clinic, San Francisco, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Comprehensive Neuroscience, Inc., St. Petersburg, Florida
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Michigan Head-Pain and Neurological Institute, Ann Arbor, Michigan
  - Headache Care Center/Clinvest, Springfield, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Regional Clinical Research, Inc., Endwell, New York
  - Elkind Headache Center, Mount Vernon, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - Headache Wellness Center, Greensboro, North Carolina
  - Coastal Carolina Research Center, Inc, Mt. Pleasant, South Carolina
  - Advanced Clinical Research, Inc., West Jordan, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Screened: 17 June 2009 Last Patient: 17 December 2009
Pre-assignment Details: Subjects meeting eligibility requirements at Screening were randomized at Visit 1 to NXN-188 600 mg, sumatriptan 100 mg or placebo in a 1:1:1 ratio. Randomized subjects were instructed to take study drug when they experienced a mild to moderate migraine headache with aura. Sunbjects not meeting the dosing criteria were discontinued from the study.
Groups:
- Placebo: 3 x 0 mg capsules
- NXN-188 600 mg: 3 x 200 mg capsules
- Sumatriptan Succinate 100 mg: 1 x 100 mg, 2 x 0 mg capsules
Period: Overall Study
Arm/Group | Placebo | NXN-188 600 mg | Sumatriptan Succinate 100 mg
Started | 82 | 82 | 75
Completed | 63 | 60 | 62
Not Completed | 19 | 22 | 13
Not completed — Lost to Follow-up | 2 | 3 | 1
Not completed — Study drug dosing criteria not met | 17 | 19 | 12

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | NXN-188 600 mg | Sumatriptan Succinate 100 mg | Total
Number analyzed (Participants) | 63 | 60 | 62 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] — Safety Population - included all subjects who were randomized and dosed with study drug.
  years | 37.2 (10.90) | 41.4 (13.02) | 41.2 (12.03) | 39.9 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Population - included all subjects who were randomized and dosed with study drug.
  Participants
    Female | 43 | 49 | 9 | 101
    Male | 20 | 11 | 53 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Safety Population - included all subjects who were randomized and dosed with study drug.
  Participants
    Hispanic or Latino | 3 | 6 | 3 | 12
    Not Hispanic or Latino | 60 | 54 | 59 | 173
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Safety Population - included all subjects who were randomized and dosed with study drug.
  Participants
    American Indian or Alaska Native | 1 | 0 | 0 | 1
    Asian | 0 | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
    Black or African American | 9 | 10 | 8 | 27
    White | 53 | 47 | 54 | 154
    More than one race | 0 | 1 | 0 | 1
    Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] — Safety Population - included all subjects who were randomized and dosed with study drug.
  kg | 76.6 (16.95) | 76.3 (16.61) | 74.2 (14.50) | 75.7 (16.00)
Height [Mean (Standard Deviation); unit: cm] — Safety Population - included all subjects who were randomized and dosed with study drug.
  cm | 169.5 (9.01) | 167.8 (8.67) | 166.3 (8.82) | 167.9 (8.89)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Safety Population - included all subjects who were randomized and dosed with study drug.
  kg/m^2 | 26.5 (4.54) | 27.0 (5.31) | 26.9 (4.48) | 26.8 (4.76)
Applicable Aura Symptoms for Qualifying Migraine [Number; unit: Participants] — Safety Population - included all subjects who were randomized and dosed with study drug.
  Subject may have reported more than one aura symptom.
  Participants
    Flickering lights | 33 | 40 | 39 | 112
    Spots | 43 | 43 | 43 | 129
    Lines | 13 | 12 | 11 | 36
    Loss of Vision | 22 | 18 | 22 | 62
    Pins and needles | 11 | 15 | 9 | 35
    Numbness | 7 | 10 | 11 | 28
    Dysphasia (speech disturbance) | 7 | 6 | 7 | 20
Type of Migraine [Number; unit: Participants] — Subjects are counted once within each type where at least one migraine is recorded.
  Participants
    Without Aura | 35 | 31 | 29 | 95
    With Aura | 61 | 59 | 62 | 182
Number of Previous Migraines per month [Mean (Standard Deviation); unit: migraines per month] — Number of Previous Migraines for each subject was based on the total number of migraine entries reported on the Migraine History CRF.
  migraines per month | 1.6 (0.59) | 1.5 (0.50) | 1.5 (0.50) | 1.5 (0.53)

OUTCOME MEASURES:

1. Primary Outcome: Time (Hours) to First Use of Rescue Medication
Time Frame: 24 hours
Population: The Full Analysis Set included all those subjects randomized who had dosed with study drug and had at least one (1) post study drug administration observation for headache severity. The Efficacy Evaluable Analysis Set, included all subjects with an imputed (LOCF) HSS at both the 2 hour time point and the 4 hour time point.
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Placebo: Three capsules containing placebo
- NXN-188: 600 mg of NXN-188 provided as 3 x 200 mg capsules.
- Sumatriptan Succinate: 100 mg of sumatriptan succinate provided as 1 capsule containing 100 mg of sumatriptan and 2 capsules containing placebo
Arm/Group | Placebo | NXN-188 | Sumatriptan Succinate
Number analyzed (Participants) | 63 | 60 | 62
hours | NA [10.1 to NA] — The median time to rescue was not estimable by Kaplan-Meier because an insufficient number of subjects took rescue medication in this data set for any dose group. | NA [6.4 to NA] — The median time to rescue was not estimable by Kaplan-Meier because an insufficient number of subjects took rescue medication in this data set for any dose group. | NA [NA to NA] — The median time to rescue was not estimable by Kaplan-Meier because an insufficient number of subjects took rescue medication in this data set for any dose group.
Statistical Analysis 1: Comparison: Placebo vs NXN-188; Test type: Superiority or Other; p = 0.6407, Log Rank

2. Secondary Outcome: Headache Relief and Recurrence (Observed Cases)
Description: Headache relief is defined as a ≥ 1-point reduction from baseline in Headache Severity Score. The Headache Severity Score is a four-point scale: 0=no pain; 1 = mild pain; 2 = moderate pain; and 3 = severe pain.
  Headache recurrence is defined as any subject that experiences headache relief within 4 hours, who did not use rescue medication, and who experienced a worsening of their headache to moderate or severe within 24 hours following study drug administration.
Time Frame: 2, 4 and up to 24 hours
Population: Number of subjects who experienced headache relief within 4 hours
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | NXN-188 600 mg | Sumatriptan Succinate 100 mg
Number analyzed (Participants) | 60 | 62 | 63
percentage of participants
  Headache Relief - 2 hours | 59.6 | 62.0 | 69.1
  Headache Relief - 4 hours | 73.5 | 81.1 | 81.8
  Headache Recurrence | 5.6 | 11.1 | 13.9

3. Secondary Outcome: 2 Hours Post Administration - Incidence of Complete Headache Relief, Photophobia, Phonophobia and Nausea
Description: Complete headache relief is defined as reduction of headache severity from moderate or severe to absent.
  Presence of Photophobia and Phonophobia measured on a 2-point scale: 0 = absent; 1 = present
  Nausea was measured on a 4-point scale: 0 = no nausea; 1 = mild nausea; 2 = moderate nausea; 3 = severe nausea
Time Frame: 2 hours
Population: Number of subjects with headache relief at 2 hours.
Measure: Number; unit: Participants
Arm/Group | Placebo | NXN-188 600 mg | Sumatriptan Succinate 100 mg
Number analyzed (Participants) | 47 | 50 | 55
Participants
  Complete Headache Relief-Observed Cases | 12 | 6 | 12
  Photophobia-Shift from Baseline (present-absent) | 16 | 14 | 30
  Phonophobia-Shift from Baseline (present-absent) | 18 | 30 | 22
  Nausea Score-Improvement from Baseline | 18 | 17 | 23

4. Secondary Outcome: 4 Hours Post Administration - Incidence of Complete Headache Relief, Photophobia, Phonophobia and Nausea
Description: as for outcome 3
Time Frame: 4 hours
Population: Number of subjects with headache relief at 4 hours.
Measure: Number; unit: Participants
Arm/Group | Placebo | NXN-188 600 mg | Sumatriptan Succinate 100 mg
Number analyzed (Participants) | 49 | 43 | 44
Participants
  Complete Headache Relief-Observed Cases | 21 | 19 | 22
  Photophobia-Shift from Baseline (present-absent) | 31 | 29 | 30
  Phonophobia-Shift from Baseline (present-absent) | 25 | 25 | 21
  Nausea Score-Improvement from Baseline | 23 | 26 | 29

5. Secondary Outcome: 24 Hours Post Administration - Incidence of Complete Headache Relief, Photophobia, Phonophobia and Nausea
Description: as for outcome 3
Time Frame: 24 hours
Population: Number of subjects with headache relief at 24 hours.
Measure: Number; unit: Participants
Groups:
- Sumatriptan Succinate: 1 x 100 mg, 2 x 0 mg capsules
Arm/Group | Placebo | NXN-188 600 mg | Sumatriptan Succinate
Number analyzed (Participants) | 62 | 56 | 58
Participants
  Complete Headache Relief-Observed Cases | 37 | 35 | 38
  Photophobia-Shift from Baseline (present-absent) | 51 | 49 | 48
  Phonophobia-Shift from Baseline (present-absent) | 47 | 41 | 38
  Nausea Score-Improvement from Baseline | 39 | 40 | 44
  Overall Eval-Study Medication-(Good/Excellent) | 24 | 30 | 35

ADVERSE EVENTS:
Time Frame: AE data were collected beginning at Randomization until 30 days after study drug administration.
Groups:
- Placebo: Three placebo capsules were provided. All capsules were taken at the same time.
- NXN-188: 600 mg NXN-188. Three capsules each containing 200 mg of NXN-188 were provided. All capsules were taken at the same time.
- Sumatriptan Succinate: 100 mg sumatriptan. Three capsules, one containing 100 mg sumatriptan succinate and two placebo-containing capsules were provided. All capsules were taken at the same time.
Arm/Group | Placebo | NXN-188 | Sumatriptan Succinate
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/60 | 0/62
Other Adverse Events (participants affected / at risk) | 16/63 | 17/60 | 13/62
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=63) | NXN-188 (N=60) | Sumatriptan Succinate (N=62)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 8 (8)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Hyperacusis (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor may request the Investigator or Institution not to publish or disclose information related to the clinical study.